CLINICAL TRIAL: NCT04461548
Title: Micro-interventions Aiming to Optimize Expectations or Self-compassiong and Their Differential Effects
Brief Title: Micro-interventions Aiming to Optimize Expectations or Self-compassion to Improve Well-being/Reduce Stress and Their Differential Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Micro_expect_compass
Record Dates: First submitted 2020-06-23; First posted 2020-07-08 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: no Specific Clincal Condition Required (Focus is on Persons Who Are Feeling Stressed or Want to Improve Their Wellbeing)

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group 1: Best Possible Self (Experimental): Participants are asked to think and write about their best possible future self and to imagine this positive future subsequently.
  Interventions: Behavioral: Thinking, writing and imagining
- Experimental group 2: Best Possible Self + next steps (Experimental): Participants are asked to think and write about their best possible future self and what the next steps could be to reach that best possible future. Subsequently, participants are asked to imagine this positive future.
  Interventions: Behavioral: Thinking, writing and imagining
- Experimental group 3: Self-compassion (Experimental): Participants are asked to think and write about a self-compassion exercise and to imagine this content subsequently.
  Interventions: Behavioral: Thinking, writing and imagining
- Active control group (Active Comparator): Participants are asked to think and write about a neutral task that is comparable to the experimental groups.
  Interventions: Behavioral: Thinking, writing and imagining

INTERVENTIONS:
Behavioral: Thinking, writing and imagining — All participants are asked to take some time to think and write about the content of the respective intervention group. After the writing exercise (approx. 15-20 min) participants are asked to imagine that content for about 5 minutes.

SUMMARY:
The study's aim is to determine whether brief interventions (micro-interventions) aiming to optimize expectations or enhancing feelings of self-compassion are able to improve well-being/reduce perceived stress in comparison to an active control group in an online-study

DETAILED DESCRIPTION:
In this study we use a pre-post-test design to compare the effects of the (classic) best possible self intervention vs. the best possible self intervention (including ways on how to reach the imagined best possible future) vs. a self-compassion intervention vs. an active control group. We are interested in the differential effects and examine several moderators.

ELIGIBILITY:
Inclusion Criteria:

* fluent in German language
* access to a computer/tablet/smartphone with audio output/headphones

Exclusion Criteria:

* not willing to take part in an online-intervention (duration: 60 minutes)
* no access to a computer/tablet/smartphone with audio output/headphones

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
Change in perceived stress ratings | Change from pre (baseline) to post scores (approx. 30 minutes later)
  Participants are asked to rate how stressed they feel at the moment at two time points (baseline and the intervention) on a questionnaire (VAS: item ranges from 0 (not stressed at all) - 100 (very stressed). Change scores are calculated (post- minus pre-scores; pre-scores will be used as a covariate).
  e.g.Lesage, F.-X., Berjot, S., & Deschamps, F. (2012). Clinical stress assessment using a visual ana-logue scale. Occupational Medicine, 62(8), 600-605. https://doi.org/10.1093/occmed/kqs140

SECONDARY OUTCOMES:
Change in perceived (stress) burden ratings (resulting from perceived stress) | Change from pre (baseline) to post scores (approx. 30 minutes later)
  Participants are asked to rate how burdened they feel at the moment at two time points (baseline and the intervention) due to the experienced stress on a questionnaire (VAS: item ranges from 0 (not at all) - 100 (very much). Change scores are calculated (post- minus pre-scores; pre-scores will be used as a covariate). Indirect/opposite measure of well-being.
Change in emotions (PANAS) | Change from pre (baseline) to post scores (approx. 30 minutes later)
  Change scores are calculated for positive and negative sum scores (post- minus pre-scores; pre-scores will be used as a covariate).
  Krohne, H.W., Egloff, B., Kohlmann, C.W., & Tausch, A. (1996). Experiments with a German version of the "Positive and Negative Affect Schedule (PANAS). Diagnostica, 42, 139-156.
Change in state optimism ratings | Change from pre (baseline) to post scores (approx. 30 minutes later)
  State Optimism measure (SOM), 7 items (each item 1(strongly disagree)-5(strongly agree)). Change scores are calculated for positive and negative sum scores (post- minus pre-scores; pre-scores will be used as a covariate). Millstein, R. A., Chung, W. J., Hoeppner, B. B., Boehm, J. K., Legler, S. R., Mastromauro, C. A., & Huffman, J. C. (2019). Development of the State Optimism Measure. General hospital psychiatry, 58, 83-93
Change in state self-compassion | Change from pre (baseline) to post scores (approx. 30 minutes later)
  Change in state self-compassion (SCS-state), 16 items (each item 1(strongly disagree) - 5 (strongly agree)). Change scores are calculated (post- minus pre-scores; pre-scores will be used as a covariate).
  Breines, J. G., & Chen, S. (2013). Activating the inner caregiver: The role of support-giving schemas in increasing state self-compassion. Journal of Experimental Social Psychology, 49(1), 58-64. https://doi.org/10.1016/j.jesp.2012.07.015
Satisfaction ratings with the respective intervention | Only Post-Assessment (end of the experiment; approx. 45-60 minutes after start of the experiment)
  e.g. "I was satisfied with the intervention" or "I feel like I had a benefit from this intervention"
Ratings directly assessing the perceived change due to the intervention | Only Post-Assessment (end of the experiment; approx. 45-60 minutes after start of the experiment)
  e.g. "The intervention reduced my perceived stress", "The intervention increased my feeling of being able to influence things"
Change in perceived self-efficacy (expectations) | Change from pre (baseline) to post scores (approx. 30 minutes later)
  Change in perceived self-efficacy (SWE), 10 items (each item (1(not at all) - 4(exactly)). Change scores are calculated (post- minus pre-scores; pre-scores will be used as a covariate).
  SchwarzerR& Jerusalem M. Generalized Self---Efficacy scale. In J. Weinman, S. Wright, &M. Johnston, Measures in health psychology: A user's portfolio. Causal andcontrol beliefs (pp. 35---37). 1995. Windsor, England: NFER---NELSON.
Change in anxiety and depression state (STADI) | Change from pre (baseline) to post scores (approx. 30 minutes later)
  Change in anxiety and depression state (STADI), 20 items (each item 1(strongly disagree) - 4 (strongly agree)). Change scores are calculated (post- minus pre-scores; pre-scores will be used as a covariate).
  Laux, L., Hock, M., Bergner-Köther, R., Hodapp, V., & Renner, K. H. (2013). The State-Trait-Anxiety-Depression-Inventory-Manual. Göttingen, Germany: Hogrefe.

CONTACTS AND LOCATIONS:
Locations (1):
- Philipps University Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided